CLINICAL TRIAL: NCT01239641
Title: Safety and Efficacy of High Intensity Focused Ultrasound Ablation Compared With Myomectomy in Uterine Fibroids:A Randomized Controlled Study
Brief Title: High Intensity Focused Ultrasound Ablation Virus Myomectomy to Treat Uterine Fibroids
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: ZB Wang, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2610; 30901234 (Other Grant/Funding Number: Nature Science Foundation of China)
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Uterine Fibroid
Keywords: Uterine Fibroids; Myoectomy; High Intensity Focused Ultrasound; ablation
MeSH Terms: conditions — Leiomyoma | interventions — Uterine Myomectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: High intensity focused ultrasound — The term 'high intensity focused ultrasound' means using ultrasound to causes coagulation necrosis to destroy the targeted tissue, in this case, uterine fibroids.
  Other Names: myomectomy

SUMMARY:
The purpose of this study is to determine whether HIFU has superiority over traditional surgery on satisfaction and adverse impact.

DETAILED DESCRIPTION:
Uterine fibroids (leiomyomas) are common in reproductive aged women. Patients are seeking new ways to treat symptomatic uterine fibroids that allow them to avoid surgery. High intensity focused ultrasound therapy (HIFU) is a novel non-invasive method for uterine fibroid. Preliminary clinical studies proved HIFU ablation is a safe and effective technology. However, it is not clear whether HIFU has superiority over traditional surgery on satisfaction and adverse impact.The study is to confirm these questions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45; The size of fibroid situated at anterior wall not lower than 2 cm in MRI feature; The size of fibroid situated at posterior wall not lower than 4 cm in MRI feature.

Exclusion Criteria:

* Cervical fibroids; Subserosal fibroids with pedicle, the width of pedicle≤ 2cm; Type 0 submucosal fibroids according to European Gynecologic Endoscopy classification; Combined with acute reproductive inflammation, or other benign and malignant gynecological diseases such as endometriosis, ovarian cancer; Pregnant (pregnancy test is positive), and lactating women; Allergy to MRI contrast agent; The history of collagen connective tissue, radiotherapy, especially abdominal radiotherapy; Surgical and anesthetic contraindications such as serious cardiac, vascular and other systemic diseases; Poor compliance; Patients who are not subject to experimental design.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The quality of life, adverse events | 1 year

SECONDARY OUTCOMES:
Fibroid volume ablated | any time
  Detection of serum markers of trauma, The change of immunological function,Procedure duration, Time to return to normal activity ,Recurrence, Reintevention rate and Pregnancy outcome, Female reproductive function, Sexual function and psychological change

CONTACTS AND LOCATIONS:
Overall Officials: LD Tang, PhD, Study Chair — the first affiliated Chongqing University Hospital, Dept of Obstetrics and Gynecolog; Z B wang, PhD, Study Director — Biomedical Engineering Department of Chongqing Medical University; Wen-Zhi Chen, MD, Principal Investigator — Clinical Center for Tumor Therapy, the 2nd Hospital of Chongqing Medical University; Jin-Yun Chen, PhD, Principal Investigator — Biomedical Engineering Department of Chongqing Medical University; Min Zhou, PhD, Principal Investigator — The first affiliated Chongqing University Hospital, Dept of Obstetrics and Gynecology; Juan Qin, PhD, Principal Investigator — Biomedical Engineering Department, Chongqing Medical University; Xiaoyan Wang, PhD, Principal Investigator — The first affiliated Chongqing University Hospital, Dept of Obstetrics and Gynecology
Locations (1):
- The 1st Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Wang X, Qin J, Wang L, Chen J, Chen W, Tang L. Effect of high-intensity focused ultrasound on sexual function in the treatment of uterine fibroids: comparison to conventional myomectomy. Arch Gynecol Obstet. 2013 Oct;288(4):851-8. doi: 10.1007/s00404-013-2775-2. Epub 2013 Apr 7. PMID 23564052